CLINICAL TRIAL: NCT02250274
Title: Prospective Randomized Study of Immune Response to Licensed Influenza Vaccines in Children and Adolescents
Brief Title: Randomized Study of Immune Response to Licensed Influenza Vaccines in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marshfield Clinic Research Foundation (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Edward Belongia, Director of Center for Clinical Epidemiology and Population Health, Marshfield Clinic Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5U01IP000471-04 (NIH)
Record Dates: First submitted 2014-09-17; First posted 2014-09-26 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Immune Response to Influenza Vaccine; Influenza A Virus Infection; Influenza B Virus Infection
Keywords: Immune response to influenza vaccine; PCR confirmed Influenza A virus; PCR confirmed Influenza B virus
MeSH Terms: interventions — FluMist; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAIV 2014-15 (Other): Will receive LAIV this year. Includes 5-8 year olds and approximately half of the 9-17 year olds. Prior history includes vaccine failures, vaccinated/uninfected and unvaccinated/uninfected last year. PBMC available for those who were infected last year, all ages.
  Interventions: Biological: LAIV
- IIV 2014-15 (Other): Will receive IIV this year. Includes only 9-17 year olds (unless shortages of LAIV encountered). Prior history includes vaccine failures, vaccinated/uninfected and unvaccinated/uninfected last year. PBMC available for those who were infected last year, only 9-17 year olds.
  Interventions: Biological: IIV

INTERVENTIONS:
Biological: LAIV — Licensed and approved Live Attenuated Influenza Vaccination (LAIV) will be preferentially given to all children aged 5-8 years old as recommended by Advisory Committee on Immunization Practices. A modified randomization scheme in which every other child aged 9-17 years enrolled in the study will be given LAIV will be used. The rest of the children aged 9-17 years old will receive IIV.
  Other Names: FluMist
  Arms: LAIV 2014-15
Biological: IIV — A modified randomization scheme in which every other child aged 9-17 years enrolled in the study will be given IIV will be used. The rest of the children 9-17 years old will receive LAIV.
  [Note: Although we do not anticipate exhausting the supply of LAIV, should this occur, children aged 5-8 will be offered IIV as it is also approved in this age group and should be used if LAIV is unavailable.]
  Other Names: FluZone
  Arms: IIV 2014-15

SUMMARY:
The purpose of this study is to assess the serologic and cell-mediated immune response to licensed live attenuated influenza vaccine (LAIV) and inactivated influenza vaccine (IIV) in children 5-17 years old. The effects of prior infection and or prior season vaccination will be examined. Children will be followed during the influenza season to identify laboratory-confirmed influenza (i.e. vaccine failure).

DETAILED DESCRIPTION:
All children will have baseline blood samples drawn and will then be vaccinated with licensed and approved influenza vaccines. Following the recommendation from the Advisory Committee on Immunization Practices, children 5-8 years old will preferentially receive live attenuated influenza vaccine (LAIV). Children aged 9-17 will be randomized to receive either LAIV or inactivated influenza vaccine (IIV). Children with a medical contraindication to any licensed influenza vaccine will be excluded from the study.

The children will have their blood drawn between 2 and 4 times total over the course of two months in order to test their immune response to the vaccine. Between approximately December and April, study participants will be contacted weekly to monitor for any new respiratory illnesses with cough, and if present, nasal and throat swabs will be collected to test for influenza.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-17 years for the duration of the study period (Sept 1, 2014-Apr 1, 2015)
* Enrolled in either the immune response study or the vaccine effectiveness study conducted at the site in the 2013-14 influenza season
* If enrolled in the vaccine effectiveness study the previous season must have either been vaccinated and infected with influenza or unvaccinated and uninfected with influenza

Exclusion Criteria:

* Children with contraindications to either the quadrivalent live attenuated influenza vaccine or to the trivalent inactivated influenza vaccine will be excluded.
* Anyone unwilling or unable to complete all required study activities including informed consent
* Subjects who already received the influenza vaccine for the 2014-15 season

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Belongia, MD, Principal Investigator — Marshfield Clinic Research Foundation - Center for Clinical Epidemiology & Population Health
Locations (1):
- Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is a plan to publish the results of the study in a manuscript but no plans to release individual level data as the results are not clinically actionable.

RESULTS

PARTICIPANT FLOW:
Groups:
- IIV 2014-15: Will receive IIV this year. Includes only 9-17 year olds (unless shortages of LAIV encountered). Prior history includes vaccine failures, vaccinated/uninfected and unvaccinated/uninfected last year. PBMC available for those who were infected last year, only 9-17 year olds.
  IIV: A modified randomization scheme in which every other child aged 9-17 years enrolled in the study will be given IIV will be used. The rest of the children 9-17 years old will receive LAIV.
  [Note: Although we do not anticipate exhausting the supply of LAIV, should this occur, children aged 5-8 will be offered IIV as it is also approved in this age group and should be used if LAIV is unavailable.]
Period: Overall Study
Arm/Group | LAIV 2014-15 | IIV 2014-15
Started | 85 | 46
Completed | 78 | 40
Not Completed | 7 | 6
Not completed — Insufficient blood draw amount | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAIV 2014-15 | IIV 2014-15 | Total
Number analyzed (Participants) | 85 | 46 | 131
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 10 (3.2) | 12 (2.5) | 11 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 21 | 56
  Male | 50 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Titer Response to Vaccine and Circulating Strains of Influenza
Time Frame: Change from Baseline to 28 days
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | LAIV 2014-15 | IIV 2014-15
Number analyzed (Participants) | 78 | 40
Titers
  H3N2 Day 28 HI Titer | 99 [79 to 124] | 295 [227 to 383]
  H3N2 Baseline HI Titer | 96 [76 to 122] | 100 [67 to 149]

2. Secondary Outcome: Polymerase Chain Reaction (PCR) Confirmed Influenza Illness
Time Frame: Onset >13 days after vaccination and before April 1, 2015
Measure: Number; unit: participants
Arm/Group | LAIV 2014-15 | IIV 2014-15
Number analyzed (Participants) | 85 | 46
participants | 13 | 5

3. Secondary Outcome: Antibody Dependent Cellular Cytotoxicity (ADCC) Titers
Time Frame: Change from Baseline to 28 days
Population: Fold change in NK cell degranulation
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Groups:
- IIV-IIV: Participants receiving IIV in 2013-14 and IIV again in 2014-15.
- IIV-LAIV: Participants receiving IIV in 2013-14 and LAIV in 2014-15.
- LAIV-IIV: Participants receiving LAIV in 2013-14 and IIV in 2014-15.
- LAIV-LAIV: Participants receiving LAIV in 2013-14 and LAIV in 2014-15.
- Unvax-IIV: Participants unvaccinated in 2013-14 and receiving IIV in 2014-15.
- Unvax-LAIV: Participants unvaccinated in 2013-14 and receiving LAIV in 2014-15.
Arm/Group | IIV-IIV | IIV-LAIV | LAIV-IIV | LAIV-LAIV | Unvax-IIV | Unvax-LAIV
Number analyzed (Participants) | 19 | 31 | 13 | 28 | 7 | 10
Fold change
  Fold change in NK cell degranulation to SW antigen | 1.02 [0.76 to 1.36] | 0.99 [0.93 to 1.05] | 1.47 [1.03 to 2.09] | 0.86 [0.76 to 0.98] | 1.31 [0.96 to 1.8] | 1.08 [0.90 to 1.29]
  Fold change in NK cell degranulation to TX antigen | 1.10 [0.96 to 1.25] | 0.95 [0.86 to 1.06] | 1.39 [1.18 to 1.64] | 1.01 [0.92 to 1.11] | 1.13 [0.75 to 1.70] | 1.33 [1.18 to 1.49]

4. Secondary Outcome: Ratio Between Immunoglobulin A (IgA):Immunoglobulin G (IgG)
Time Frame: Day 7
Population: There were too few samples collected within each group to conduct a reasonable analysis of this outcome. The samples collected are being stored for potential future use.
Arm/Group | LAIV 2014-15 | IIV 2014-15
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | LAIV 2014-15 | IIV 2014-15
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/46
Other Adverse Events (participants affected / at risk) | 0/85 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No